CLINICAL TRIAL: NCT01052948
Title: The Association Between Dopamine Agonists and Cardiac Valvulopathy, Fibrosis and Other Cardiopulmonary Events
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Other Study IDs: A7231031
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Results first posted 2011-03-11 (Estimated); Last update posted 2011-03-23 (Estimated); Status verified 2011-03

CONDITIONS: Parkinson's Disease; Hyperprolactinemia
Keywords: dopamine agonists; cabergoline; Parkinson's disease; hyperprolactinemia; epidemiology; cardiac valvulopathy
MeSH Terms: conditions — Parkinson Disease; Hyperprolactinemia; Heart Valve Diseases | interventions — Retrospective Studies

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- Cohort 1: All persons who newly start one of the dopamine agonists (DA) after start of eligibility period
  Interventions: Other: Retrospective study-
- Cohort 2: All persons who started levodopa after start of eligibility period and had not been treated with dopamine agonists anytime prior.
  Interventions: Other: Retrospective study-
- Cohort 3: All persons with newly diagnosed hyperprolactinemia who had not been treated with dopamine agonists anytime prior.
  Interventions: Other: Retrospective study-
- Cohort 4: healthy controls from general population matched on age, gender, index date and general practitioner (GP) practice to persons exposed to dopamine agonists
  Interventions: Other: Retrospective study-

INTERVENTIONS:
Other: Retrospective study-
  Groups: Cohort 1
Other: Retrospective study-
  Groups: Cohort 2
Other: Retrospective study-
  Groups: Cohort 3
Other: Retrospective study-
  Groups: Cohort 4

SUMMARY:
To assess the association between cabergoline and other dopamine agonists (DAs), and symptomatic, diagnosed serious cardiopulmonary disorders, including:

1. Cardiac valve regurgitation
2. Diffuse Pleural/pulmonary thickening and pericardial and retroperitoneal fibrosis
3. Heart failure
4. Total, cardiac and respiratory mortality

ELIGIBILITY:
Inclusion Criteria:

* At least one year registered with the general practitioner (GP), one year of valid data from the GP, or the date of software conversion (if GP software systems had changed) and meeting criteria for any one of the 4 cohorts as defined.

Exclusion Criteria:

* rheumatic heart disease
* congenital heart disease: includes structural defects, congenital arrhythmias, and cardiomyopathies
* dilated cardiomyopathy (congestive cardiomyopathy
* pericardial, pleural, pulmonary or retroperitoneal fibrosis
* endocarditis or myocarditis
* carcinoid syndrome
* intravenous drug abuse
* fibrotic valvular heart disease
* pleural/pulmonary/pericardial/retroperitoneal fibroses
* use of fenfluramine or amiodarone within 3 years prior to date of diagnosis of fibrotic valvular heart disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: General research practice databases or record linkage systems in Europe that provide access to original medical information. These are: The Health Information Network (THIN), Health Search Database (HSD)-THALES, the Integrated Primary Care Information (IPCI) and PHARMO-Record Linkage System (RLS) and meeting criteria for entry into any of the 4 cohorts between 1995 - 2007
Sampling Method: Non-Probability Sample
Enrollment: 86939 (Actual)
Dates: Start 2007-01; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A7231031&StudyName=The%20Association%20between%20Dopamine%20Agonists%20and%20Cardiac%20Valvulopathy%2C%20Fibrosis%20and%20Other%20Cardiopulmonary%20Events

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Noninterventional retrospective cohort study.
Groups:
- Dopamine Agonist (Cohort 1): Participants with Parkinson's Disease (PD)/Parkinsonism, Restless Legs Syndrome (RLS) or hyperprolactinemia (previously treated) who newly started one of the ergot-derived Dopamine Agonists (DAs): Lisuride, Cabergoline, Metergoline, Bromocriptine, Pergolide, Dihydroergocryptine mesylate, Quinagolide, Ropinirole, Pramipexole, Piribedil, or Rotigotine.
- Levodopa (Cohort 2): Participants with PD/Parkinsonism or RLS who newly started treatment with Levodopa: Levodopa and decarboxylase inhibitor; Levodopa, decarboxylase inhibitor and catechol-O-methyl transferase [COMT] inhibitor; MeLevodopa; MeLevodopa and decarboxylase inhibitor; or EtiLevodopa and decarboxylase inhibitor and had not been treated with DAs anytime prior.
- Hyperprolactinemia (Cohort 3): Participants with newly diagnosed hyperprolactinemia (excluding postpartum hyperprolactinemia), who had not been treated with DAs anytime prior.
- Healthy Controls (Cohort 4): Healthy control participants matched (1:1) with participants in the DA cohort (Cohort 1) for age (exact year), gender, database and date of start of DA.
Period: Overall Study
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4)
Started | 27812 | 14669 | 15147 | 29311
Completed | 27812 | 14669 | 15147 | 29311
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4) | Total
Number analyzed (Participants) | 27812 | 14669 | 15147 | 29311 | 86939
Age Continuous [Mean (Standard Deviation); unit: years] | 48.7 (20.1) | 76.8 (0.1) | 40.0 (0.1) | 49.4 (0.1) | 52.0 (21.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22084 | 7666 | 13398 | 21992 | 65140
  Male | 5728 | 7003 | 1749 | 7319 | 21799

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Fibrotic Valvular Heart Disease Per 10,000 Participant-Years of Follow-Up
Description: Occurrence of: mitral stenosis with insufficiency, other unspecified mitral valve diseases, mitral or aortic valve stenosis, insufficiency, or disorders, multiple involvement of mitral and aortic valves, mitral and aortic valve diseases, unspecified, diseases of tricuspid valve, tricuspid valve disorders, specified as nonrheumatic, pulmonary valve disorders, endocarditis, valve unspecified, endomyocardial fibrosis, endocardial fibroelastosis, other primary or secondary cardiomyopathies, cardiomyopathy, functional and undiagnosed cardiac murmurs, other abnormal heart sounds.
Time Frame: Up to 12 years
Population: Per protocol.
Measure: Number; unit: Participants/10,000 Participant-Years
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4)
Number analyzed (Participants) | 27812 | 14669 | 15147 | 29311
Participants/10,000 Participant-Years | 21 | 21 | NA — Due to limited number of exposed cases in hyperprolactinemia cohort, no additional analyses beyond exploration of cabergoline and other single products (current, past) vs non-use, and where possible, dose/duration effect could be performed. | 52

2. Primary Outcome: Number of Participants With Fibrosis Per 10,000 Participant-Years of Follow-Up
Description: Occurrence of: idiopathic retroperitoneal fibrosis, occlusion not otherwise specified (NOS) of ureter, diffuse (idiopathic) (interstitial) pulmonary fibrosis, Hamman-Rich syndrome, interstitial pneumonia (desquamative) (lymphoid), fibrosis of lung (atrophic; confluent; massive; perialveolar; peribronchial) chronic or unspecified, pulmonary or pleural fibrosis, abnormal communication between pericardial and pleural sacs, pleural fold anomaly, adhesive or constrictive pericarditis, pericardial fibrosis
Time Frame: Up to 12 years
Population: Per protocol.
Measure: Number; unit: Participants/10,000 Participant-Years
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4)
Number analyzed (Participants) | 27812 | 14669 | 15147 | 29311
Participants/10,000 Participant-Years | 2 | 5 | NA — Due to limited number of exposed cases in hyperprolactinemia cohort, no additional analyses beyond exploration of cabergoline and other single products (current, past) vs non-use, and where possible, dose/duration effect could be performed. | 8

3. Primary Outcome: Number of Participants With Heart Failure Per 10,000 Participant-Years of Follow-Up
Description: Occurrence of: unspecified acute edema of lung, heart failure, acute pulmonary heart disease, or acute cor pulmonale
Time Frame: Up to 12 years
Population: Per protocol.
Measure: Number; unit: Participants/10,000 Participant-Years
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4)
Number analyzed (Participants) | 27812 | 14669 | 15147 | 29311
Participants/10,000 Participant-Years | 69 | 161 | NA — Due to limited number of exposed cases in hyperprolactinemia cohort, no additional analyses beyond exploration of cabergoline and other single products (current, past) vs non-use, and where possible, dose/duration effect could be performed. | 201

4. Primary Outcome: Number of Participants With All-Cause Mortality Per 10,000 Participant-Years of Follow-Up
Description: All participants who died independent of the cause to include instantaneous death, death occurring in less than 24 hours from onset of symptoms, not otherwise explained, unattended death and other causes of ill defined morbidity and mortality. Cause of death was coded and classified as either cardiovascular or respiratory.
Time Frame: Up to 12 years
Population: Per protocol.
Measure: Number; unit: Participants/10,000 Participant-Years
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4)
Number analyzed (Participants) | 27812 | 14669 | 15147 | 29311
Participants/10,000 Participant-Years | 170 | 803 | NA — Due to limited number of exposed cases in hyperprolactinemia cohort, no additional analyses beyond exploration of cabergoline and other single products (current, past) vs non-use, and where possible, dose/duration effect could be performed. | 719

ADVERSE EVENTS:
Description: Information about adverse events was not collected during this observational, noninterventional, case control study.
Arm/Group | Dopamine Agonist (Cohort 1) | Levodopa (Cohort 2) | Hyperprolactinemia (Cohort 3) | Healthy Controls (Cohort 4)
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.